CLINICAL TRIAL: NCT06997471
Title: A Phase I, Single-Center, Open-Label Trial to Assess the Safety and Tolerability of Delayed Infusion of a Naïve T Cell Depleted Hematopoietic Graft and Memory T-lymphocytes in Recipients of Solid Organ Transplantation
Brief Title: Phase I Trial on the Safety of Delayed Infusion of a Naïve T Cell-Depleted Hematopoietic Graft With Memory T Cells in Solid Organ Transplant Recipients
Acronym: DUALGRAFT
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Francisco Hernández Oliveros (Other)
Responsible Party: Sponsor-Investigator, Francisco Hernández Oliveros, Physician in the Department of Pediatric Surgery. Head of the Pediatric Transplant Section., Hospital Universitario La Paz
Organization: Hospital Universitario La Paz (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DUALGRAFT
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Solid Organ Transplant Complications; Solid Organ Transplant Recipients; Solid Organ Transplant Rejection
MeSH Terms: interventions — Antigens, CD34

STUDY DESIGN:
Intervention Model Description: This study is a single-center, open-label clinical trial. Its primary goal is to evaluate the safety of inducing hematopoietic mixed chimerism to promote immunological tolerance in SOT recipients. A total of 10 participants will be recruited, either prior to their scheduled SOT or having already undergone SOT (in case of renal transplant recipients with a living donor), depending on enrollment feasibility.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSCT using a graft enriched in CD34+ hematopoietic progenitor cells (Experimental): The study intervention involves a HSCT using a graft enriched in CD34+ hematopoietic progenitor cells. This graft will be specifically engineered through depletion of naïve T-lymphocytes (CD45RA+) and patients will be supplemented with memory lymphocytes to support immune reconstitution and promote tolerance. The source of the hematopoietic stem cells (HSCs) will vary depending on whether the donor is a living related donor (HLA-identical or haploidentical) or a deceased donor.
  Graft Composition and Cell Doses
  * CD34+ cells: < 1 x 107/kg will be intravenously infused as the primary source of hematopoietic progenitors.
  * Memory T-lymphocytes (CD45RO+): < 3 x 107/kg will be administered. Naïve T-lymphocytes (CD45RA+) remaining in the memory fraction will always be <1 x 104/kg, to minimize the risk of GVHD while supporting immune surveillance.
  * Only in haploidentical participants: NK cells (CD56+): < 5 x 107/kg to promote graft tolerance and target residual malignant cells.
  Interventions: Biological: Investigational cellular therapy consisting on a HSCT using a graft enriched in CD34+, depleted of naïve T-lymphocytes and supplemented with memory lymphocytes

INTERVENTIONS:
Biological: Investigational cellular therapy consisting on a HSCT using a graft enriched in CD34+, depleted of naïve T-lymphocytes and supplemented with memory lymphocytes — Infusion Schedule
  1. Primary Infusion: the enriched graft, containing the CD34+ progenitors and depleted naïve T cells, will be infused after the patient has undergone conditioning therapy.
  2. In the case of haploidentical donors, an additional NK cell infusion will be administered whenever possible around day 7 post-transplant from a non-mobilized apheresis collection, aiming to enhance graft tolerance and prevente HHV6 disease.
  3. Post-Transplant Memory T cell Infusions: beginning on days 15 and 30, and then administered monthly up to a maximum of one year or until the supply is depleted, memory T cells will be infused.
  Conditioning Regimen
  Prior to HSCT, all patients will undergo a low-intensity conditioning regimen designed to allow engraftment of the donor cells while minimizing toxicity:
  1. Total Lymphoid Irradiation (TLI): 8 Gy of total lymphoid irradiation will be administered.
  2. Fludarabine: a total dose of 120 mg/m², spread over 4 days (-6 to -3 before transplant), will serv

SUMMARY:
The goal of this clinical trial is to evaluate the safety and feasibility of inducing hematopoietic mixed chimerism to promote immune tolerance and potentially reduce the need for lifelong immunosuppression in pediatric and adult patients undergoing solid organ transplantation (SOT), including kidney, lung, and multivisceral transplants.

The main questions it aims to answer are:

* Is it safe to infuse a naïve T cell-depleted hematopoietic graft along with memory T-lymphocytes after SOT?
* Can this approach support immune tolerance and reduce the incidence of rejection and infection without long-term immunosuppression?

Participants will:

* Undergo a solid organ transplant from a living or deceased donor.
* Wait through a stabilization period to ensure resolution of early transplant-related complications.
* Receive low-dose preconditioning (TLI and thymic irradiation) to prepare for hematopoietic stem cell transplantation.
* Be infused with a graft containing CD34+ progenitor cells, memory T cells (CD45RO+), and no naïve T cells (CD45RA+); in some cases, NK cells may also be included.
* Be followed for graft survival, immune tolerance, infection rates, and adverse events through regular clinical and immune monitoring visits.

DETAILED DESCRIPTION:
This clinical trial is exploring a new way to help patients who receive a solid organ transplant-such as a kidney, lung, or intestine-live longer and healthier lives with fewer side effects from medication. Today, most transplant recipients must take strong immune-suppressing drugs every day to prevent their bodies from rejecting the new organ. While these drugs are essential, they can lead to serious complications over time, such as infections, and even damage to the transplanted organ itself.

The goal of this study is to test a promising strategy that may help the body naturally accept the transplanted organ, reducing or potentially eliminating the need for long-term immunosuppressive drugs. This approach involves a technique called mixed hematopoietic chimerism, which means that the patient's body receives a mix of immune cells from both themselves and the organ donor. When successful, this blend of immune systems can lead to immune tolerance, allowing the transplanted organ to function without being attacked by the patient's immune system.

This is a Phase I, single-center, open-label clinical trial, which means it is an early-stage study focused primarily on evaluating safety. The trial will enroll 10 patients who are either scheduled to receive a solid organ transplant (SOT) or have recently undergone one, depending on the type of organ and donor availability.

After a transplant, each patient must go through a stabilization period, allowing time for any immediate post-surgical complications to improve. Once stabilized, the patient will receive a specially prepared infusion of blood-forming (hematopoietic) stem cells from their organ donor. This process is known as hematopoietic stem cell transplantation (HSCT).

Before this infusion, patients will undergo low-dose preconditioning using total lymphoid irradiation (TLI) and thymic irradiation. These treatments prepare the body to accept the donor's cells without causing major immune damage, and they aim to lower the risk of complications like graft-versus-host disease (GVHD)-a serious condition where donor immune cells attack the patient's tissues.

The infused cell product is carefully designed:

* It includes CD34+ blood stem cells, which help rebuild the patient's immune and blood systems.
* It removes "naïve" T cells (CD45RA+), which are known to cause GVHD.
* It includes "memory" T cells (CD45RO+), which support immune recovery and protection against infections.

In some cases, natural killer cells CD56+ may also be included to help protect against viruses and support tolerance-especially when the donor is haploidentical.

The way the cells are collected depends on whether the donor is living or deceased. For living donors, peripheral blood stem cells are collected. For deceased donors, the bone marrow is used.

This trial is based on encouraging results from earlier studies and aims to show that this strategy is safe and feasible. If successful, the benefits could be wide-ranging:

* Less dependence on lifelong immunosuppressive medications
* Lower risk of chronic rejection of the transplanted organ
* Fewer life-threatening infections
* Improved quality of life, especially for children and young adults
* Increased availability of transplantable organs by improving outcomes and reducing re-transplantation needs
* Lower healthcare costs due to fewer complications, hospitalizations, and medications

The study will also track how well the patient's body accepts the transplanted organ over time and whether true immune tolerance is achieved. This will be monitored by looking at immune markers in the blood and through regular clinical follow-ups.

This approach could be especially helpful for pediatric patients, who face unique challenges, such as difficulty adhering to lifelong medication plans and a higher risk of needing multiple transplants. It may also help adult patients at high risk of rejection, or those who have already had complications with previous transplants.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (<18 years old) who are candidates to receive intestinal or lung transplantation (before SOT).
* Pediatric (<18 years old) or adult patients (≥18 years old) who are either candidates for renal transplantation or have already undergone renal transplantation and remain candidates for subsequent HSCT.
* Patients who provide informed consent (or their legal guardians in the case of minors) before any study-related procedures.
* Recipients should have no active infectious disease or other medical condition that would contraindicate the combined transplantation procedure, as determined by the investigational team.

Exclusion Criteria:

* Recipients with existing bone marrow disorders or those receiving medications known to adversely affect bone marrow function.
* Patients with advanced organ dysfunction (hepatic, cardiac, or pulmonary) incompatible with successful combined transplantation.
* Patients with active or uncontrolled autoimmune conditions that may interfere with transplantation and the induction of chimerism.
* Patients with known allergies to medications or products required for conditioning or transplantation.
* Patients with severe psychiatric or cognitive disorders that may interfere with adherence to study instructions or postoperative care.
* Patients currently enrolled in another clinical trial that could interfere with the outcomes or safety of this study.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Any other condition that, in the opinion if the Investigator, may interfere with the efficacy and/or safety evaluation of the trial.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events related to the investigational intervention. | From enrollment to end of follow-up at 2 years after cell therapy administration
  Safety and tolerability will be evaluated based on the incidence, nature and and severity of adverse events during study period. (clinical and laboratory).

SECONDARY OUTCOMES:
Feasibility of cell collection, processing and administration. | From enrollment to 3 months after solid organ transplantation
  * Proportion (%) of participants in which we are able to obtain naïve T cell depleted graft and memory T cells, from alive and deceased donors.
  * Prorportion (%) of participants in which we are able to obtain naïve T cell depleted graft and memory T cells from deceased donors.
  * Proportion (%) of patients who are able to proceed to haematopoietic stem cell therapy within 3 months following solid organ transplantation.
Mixed hematopoietic chimerism measurement. | From therapy administration to 30 days and 100 days after investigational therapy administration
  Proportion (%) of patients presenting mixed hematopoietic chimerism ≥ 100 days, macrochimerism (>5%) ≥ 100 days, macrochimerism ≥ 30 days and microchimerism (< 5%) ≥ 30 days.
Donor-Specific T Cell Clone Depletion | One year post haematopoietic stem cell therapy and thereafter.
  Proportion (%) of patients demonstrating donor's alloreactive clones depletion by high resolution TCR sequencing one year post haematopoietic stem cell therapy and thereafter.
Organ Rejection Rate | From investigational therapy administration to 1 year after
  Proportion (%) of patients experiencing organ rejection 1 year after investigational therapy administration.
Graft Survival and Failure Rates | From enrollment to end of follow-up at 2 years after cell therapy administration
  Survival rate of grafts, rates of graft failure or complications.
occurence of GVHD in patients receiving delayed infusion of the investigational celular therapy after solid organ transplantation. | From enrollment to end of follow-up at 2 years after cell therapy administration
  Proportion (%) of patients presenting GVHD, GVHD grade 1 and GVHD garde >1
Occurrence of infections in patients receiving delayed infusion of the investigational celular therapy after solid organ transplantation. | From enrollment to end of follow-up at 2 years after cell therapy administration
  Proportion (%) of patients experiencing sepsis or requiring intensive care due to an investigational treatment related adverse event, of viral reactivations/infections, fungal disease, and bacterial infections after investigational treatment initiation.
Immune reconstitution in patients receiving delayed infusion of the investigational celular therapy after solid organ transplantation | Day 100 post haematopoietic stem cell therapy.
  Proportion (%) of patients with CD4+ count >200 cells/μL on day 100 post haematopoietic stem cell therapy.
Immune reconstitution in patients receiving investigational cell therapy | From enrollment to end of follow-up at 2 years after cell therapy administration
  Proportion (%) of patients with Treg percentage > 10% at any point after haematopoietic stem cell therapy.
Development of immune tolerance in transplant recipients | One-year post haematopoietic stem cell therapy and thereafter.
  Proportion (%) of patients demonstrating donor's alloreactive clones depletion by high resolution TCR sequencing and proportion (%) of patients experiencing organ rejection one year post haematopoietic stem cell therapy and thereafter.
Recipient's laboratory hyporesponsiveness towards the graft | One-year post haematopoietic stem cell therapy and thereafter.
  Proportion (%) of patients with donor's hyporesponsiveness in Mixed Lymphocyte Reaction (MLR) one-year post haematopoietic stem cell therapy and thereafter.
Recipient's competence against third party donors | One-year post haematopoietic stem cell therapy and thereafter.
  Proportion (%) of patients with third party response in Mixed Lymphocyte Reaction (MLR) one-year post haematopoietic stem cell therapy and thereafter.
Recipient's competence against virus | One-year post haematopoietic stem cell therapy and thereafter.
  Proportion (%) of patients with competent viral immune response in functional tests one-year post haematopoietic stem cell therapy and thereafter.
Mortality after investigational therapy adminitration. | From enrollment to one year after investigational therapy administration
  Proportion (%) of patients alive up to 1 year after investigational therapy administration.